CLINICAL TRIAL: NCT04075474
Title: Preventing Early Childhood Caries With Silver Diamine Fluoride - a Randomised Clinical Trial
Brief Title: Preventing Early Childhood Caries With Silver Diamine Fluoride
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun-Hung Chu, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW18-619
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- silver diamine fluoride (Experimental): 38% silver diamine fluoride
  Interventions: Device: silver diamine fluoride
- sodium fluoride (Active Comparator): 5% sodium fluoride
  Interventions: Device: sodium fluoride

INTERVENTIONS:
Device: silver diamine fluoride — 38% SDF on primary upper anterior teeth
  Arms: silver diamine fluoride
Device: sodium fluoride — 5% NaF on primary upper anterior teeth
  Arms: sodium fluoride

SUMMARY:
Background: Silver diamine fluoride (SDF) solution is effective in arresting early childhood caries (ECC). Previous studies suggested that it might exert a preventive effect in managing ECC. However, no well-designed clinical trial has been performed to study this topic. The aim of this randomised clinical trial is to assess whether 38% SDF is superior to 5% sodium fluoride (NaF) varnish in preventing new carious lesions in primary anterior teeth.

Methods/Design: This is a Phase II single-centre randomized, double-blind, active-controlled, parallel-group pragmatic trial. The hypothesis tested is that 38% SDF is more effective than 5% NaF in preventing new caries development in primary anterior teeth. Approximately 2,100 three-year-old kindergarten children who are generally healthy and with parental consent will be recruited. This sample size is sufficient for an appropriate statistical analysis of superiority trial with power at 80%, allowing for a 15% drop-out rate. Stratified randomization will be adopted for the intervention allocation. The intervention is either 38% SDF or 5% NaF (as positive control) therapy on primary upper anterior teeth. Dental examination followed by fluoride therapy will be conducted every six months until 30 months in kindergartens by a single examiner. The examiner, children and children's parents will be blinded to the treatment allocation. Questionnaire survey will be conducted to study the children's oral health-related behaviours and their socioeconomic backgrounds.

Discussion: The effectiveness of 38% SDF in preventing ECC remains uncertain. If the results are as anticipated, it will help change the standard of care that using 5% NaF for ECC prevention. In addition, the results will be widely available and increase adoption of SDF in other countries to reduce the global burden of ECC.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy, with parental consents

Exclusion Criteria:

* uncooperative and difficult to manage, have major systemic diseases such as porphyria, or are on long-term medication such as anti-epileptic drugs.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 730 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
caries prevention | at 30-month follow-up
  the number of sound tooth surfaces that become cavitated caries per child

CONTACTS AND LOCATIONS:
Locations (1):
- Local kindergartens, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng FM, Yan IG, Duangthip D, Lo ECM, Gao SS, Chu CH. Randomized Clinical Trial on Caries Prevention of Silver Diamine Fluoride. J Dent Res. 2025 Sep 9:220345251363837. doi: 10.1177/00220345251363837. Online ahead of print. PMID 40926346
- [Derived] Gao SS, Chen KJ, Duangthip D, Wong MCM, Lo ECM, Chu CH. Preventing early childhood caries with silver diamine fluoride: study protocol for a randomised clinical trial. Trials. 2020 Feb 4;21(1):140. doi: 10.1186/s13063-020-4088-7. PMID 32019596